CLINICAL TRIAL: NCT02866370
Title: A Randomised Phase II Study Of Nintedanib (BIBF1120) Compared To Chemotherapy in Patients With Recurrent Clear Cell Carcinoma Of The Ovary Or Endometrium
Brief Title: Study Of Nintedanib Compared To Chemotherapy in Patients With Recurrent Clear Cell Carcinoma Of The Ovary Or Endometrium
Acronym: NiCCC
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: NHS Greater Glasgow and Clyde (Other)
Collaborators: Boehringer Ingelheim (Industry); Cancer Research UK (Other); European Organisation for Research and Treatment of Cancer - EORTC (Network); Nordic Society of Gynaecological Oncology - Clinical Trials Unit (Other); ARCAGY/ GINECO GROUP (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GN12ON259 (NiCCC2013); 2013-002109-73 (EudraCT Number); ISRCTN50772895 (Registry Identifier: ISRCTN); ENGOT-GYN1 (Other: ENGOT); EORTC1212 (Other: EORTC)
Record Dates: First submitted 2016-07-22; First posted 2016-08-15 (Estimated); Last update posted 2016-08-15 (Estimated); Status verified 2016-07

CONDITIONS: Ovarian Clear Cell Carcinoma; Endometrial Clear Cell Carcinoma
MeSH Terms: interventions — nintedanib; Paclitaxel; liposomal doxorubicin; Topotecan; Carboplatin; Doxorubicin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Nintedanib (Experimental): Nintedanib (BIBF1120) 200mg twice daily PO, continuously
  Interventions: Drug: Nintedanib
- Chemotherapy (Active Comparator): Ovarian Cancer Patients:
  Paclitaxel (80mg/m2) IV Day 1, 8, 15 every 28 days Pegylated Liposomal Doxorubicin (PLD) (40mg/m2) IV every 28 days Topotecan (4mg/m2) IV Day 1, 8, 15 every 28 days
  Endometrial Cancer Patients:
  Carboplatin (AUC 5) and Paclitaxel (175mg/m2) IV every 21 days Doxorubicin IV (60mg/m2) every 21 days
  Patients will usually receive up to 6 cycles of chemotherapy. If in the opinion of the Investigator, a patient would benefit from continuing with chemotherapy beyond 6 cycles, it is acceptable to continue until progression or unacceptable toxicity. The maximal lifetime cumulative dose of doxorubicin or pegylated liposomal doxorubicin allowed is 450 mg/m2.
  Interventions: Drug: Paclitaxel; Drug: Pegylated Liposomal Doxorubicin (PLD); Drug: Topotecan; Drug: Carboplatin; Drug: Doxorubicin

INTERVENTIONS:
Drug: Nintedanib — Nintedanib (BIBF1120) 200mg twice daily PO, continuously, until progression or withdrawal from the treatment.
  Other Names: BIBF 1120; Vargatef
  Arms: Nintedanib
Drug: Paclitaxel — Ovarian Cancer Patients Paclitaxel (80mg/m2) IV Day 1, 8, 15 every 28 days* Endometrial Cancer Patients Carboplatin (AUC 5) and Paclitaxel (175mg/m2) IV every 21 days*
  * Patients will usually receive up to 6 cycles of chemotherapy. If in the opinion of the Investigator, a patient would benefit from continuing with chemotherapy beyond 6 cycles, it is acceptable to continue until progression or unacceptable toxicity.
  Arms: Chemotherapy
Drug: Pegylated Liposomal Doxorubicin (PLD) — Ovarian Cancer Patients Pegylated Liposomal Doxorubicin (PLD) (40mg/m2) IV every 28 days*
  * Patients will usually receive up to 6 cycles of chemotherapy. If in the opinion of the Investigator, a patient would benefit from continuing with chemotherapy beyond 6 cycles, it is acceptable to continue until progression or unacceptable toxicity. The maximal lifetime cumulative dose of doxorubicin or pegylated liposomal doxorubicin allowed is 450 mg/m2.
  Other Names: Caelyx
  Arms: Chemotherapy
Drug: Topotecan — Ovarian Cancer Patients Topotecan 4mg/m2 IV Day 1, 8, 15 every 28 days*
  * Patients will usually receive up to 6 cycles of chemotherapy. If in the opinion of the Investigator, a patient would benefit from continuing with chemotherapy beyond 6 cycles, it is acceptable to continue until progression or unacceptable toxicity.
  Other Names: Hycamtin
  Arms: Chemotherapy
Drug: Carboplatin — Endometrial Cancer Patients Carboplatin (AUC 5) and Paclitaxel (175mg/m2) IV every 21 days*
  * Patients will usually receive up to 6 cycles of chemotherapy. If in the opinion of the Investigator, a patient would benefit from continuing with chemotherapy beyond 6 cycles, it is acceptable to continue until progression or unacceptable toxicity.
  Arms: Chemotherapy
Drug: Doxorubicin — Endometrial Cancer Patients Doxorubicin IV 60mg/m2 every 21 days*
  * Patients will usually receive up to 6 cycles of chemotherapy. If in the opinion of the Investigator, a patient would benefit from continuing with chemotherapy beyond 6 cycles, it is acceptable to continue until progression or unacceptable toxicity. The maximal lifetime cumulative dose of doxorubicin or pegylated liposomal doxorubicin allowed is 450 mg/m2.
  Arms: Chemotherapy

SUMMARY:
The trial will recruit up to 120 patients; 90 with ovarian clear cell carcinoma and up to 30 with endometrial clear cell carcinoma. Patients will be randomised between chemotherapy and Nintedanib 200mg twice daily oral administration (PO) continuously. The primary diagnosis must be histologically confirmed and central pathological review of the presenting tumour or biopsy of relapsed disease must find at least 50% clear cell carcinoma with no serous differentiation

DETAILED DESCRIPTION:
Clear cell carcinoma (CCC) is an uncommon histotype of ovarian and a rare histotype of endometrial cancer. The prognosis for recurrent disease is poor with response rates to standard chemotherapy of <10% so there is an urgent need for novel therapies. Ovarian CCC (OCCC) is biologically different from other ovarian cancer histotypes but shares features with renal CCC, including upregulation of angiogenesis pathways. Hence inhibition of angiogenesis, which has been a successful strategy in renal CCC, may also be of benefit in OCCC and endometrial CCC (ECCC).

Nintedanib is a well-tolerated, potent, orally-available, kinase inhibitor targeting Vascular Endothelial Growth Factor (VEGFR) 1-3, Platelet Derived Growth Factor Receptor (PDGFR)α/β, and Firbroblas Gworth Factor Receptors (FGFR) 1-3. It is licensed in Europe in combination with docetaxel after first line chemotherapy for Non-Small Cell Lung Cancer (NSCLC). Importantly it also has significant activity as a single agent in renal CCC with an Overall Response Rate (ORR) of 20.3%, disease control rate of 76.% and 43% 9 month progression free survival.

Response rates (RR) of ovarian CCC to standard chemotherapy with or without platinum are poor whatever line of treatment. A number of different agents are used in recurrent CCC and, although isolated instances of response to a variety of agents have been reported, no regimen seems to offer a particular advantage. As a result the investigators do not expect to see significant differences in response rates within the chemotherapy arms of the study. Hence it is feasible to allow physicians a choice of chemotherapy from a pre-specified selection and to include patients with multiple previous relapses. Since overall and progression free survival may be shorter with successive lines of treatment, the number of previous lines of treatment will be a stratification factor. These measures should maximise recruitment of this rare tumour sub-type across different countries.

ELIGIBILITY:
Inclusion Criteria:

1. Progressive or recurrent ovarian peritoneal or fallopian tube clear cell carcinoma, or progressive or recurrent endometrial clear cell carcinoma. The primary diagnosis must be histologically confirmed and central pathological review of the presenting tumour or biopsy of relapsed disease must find at least 50% clear cell carcinoma with no serous differentiation. Progressive disease as defined by Response Evaluation Criteria in Solid Tumours (RECIST) 1.1.
2. Failure after ≥1 prior platinum containing regimen which may have been given in the adjuvant setting. For patients with ovarian clear cell carcinoma, progression must have occurred within 6 calendar months of their last platinum dose.
3. ECOG (Eastern Cooperative Oncology Group) Performance status of ≤2.
4. Life expectancy of >3 months.
5. Adequate hepatic, bone marrow coagulation and renal function

   1. Hepatic function: total bilirubin < Upper Limit of Normal (ULN); ALT and AST < 2.5 x ULN
   2. Coagulation parameters: INR (International Normalised Ratio) <2 x ULN and prothrombin time and activated partial thromboplastin time < 1.5 x ULN in the absence of therapeutic anticoagulation
   3. absolute neutrophil count (ANC) ≥ 1.5 x 109/L
   4. platelets ≥ 100 x 109L
   5. haemoglobin ≥ 9.0 g/dL
   6. proteinuria < grade 2 CTCAE (version 4)
   7. Glomerular Filtration Rate ≥40ml/min. (calculated using the Wright, Cockroft & Gault equation or measured by EDTA clearance)
6. Female and > 18 years of age.
7. Signed and dated written informed consent prior to admission to the study in accordance with International Conference on Harmonization on Good Clinical Practice (ICH-GCP) guidelines and local legislation.
8. Willingness and ability to comply with scheduled visits, treatment plans and laboratory tests and other study procedures.

Exclusion Criteria:

1. Prior treatment with Nintedanib or other angiogenesis inhibitor/VEGF targeted therapy, except for prior treatment with bevacizumab which is permitted.
2. Treatment within 28 days prior to randomisation with any investigational drug, radiotherapy, immunotherapy, chemotherapy, hormonal therapy or biological therapy. Palliative radiotherapy may be permitted for symptomatic control of pain from bone metastases in extremities, provided that the radiotherapy does not affect target lesions, and the reason for the radiotherapy does not reflect progressive disease.
3. Previous treatment with the chemotherapy regimen selected as the control arm by the investigator. (Prior therapy with paclitaxel given on a three weekly regimen is permitted for patients receiving weekly paclitaxel. Prior treatment with weekly paclitaxel is permitted where this has been used as part of first line therapy and it is greater than 6 months since the last dose of weekly paclitaxel. Prior weekly paclitaxel for relapsed disease is not permitted).
4. Other malignancy diagnosed within 5 years of enrolment except for:

   1. non-melanomatous skin cancer (if adequately treated)
   2. cervical carcinoma in situ (if adequately treated)
   3. carcinoma in situ of the breast (if adequately treated)
   4. For patients with ovarian clear cell cancer, prior or synchronous endometrial cancer (if adequately treated), provided all of the following criteria are met:

      * disease stage FIGO (International Federation of Gynecology and Obstetrics) Stage 1a (tumour invades less than one half of myometrium)
      * Grade 1 or 2
5. Patients with any other severe concurrent disease, which may increase the risk associated with study participation or study drug administration and, in the judgement of the investigator, would make the patient inappropriate for entry into this study, including significant neurologic, psychiatric, infectious, hepatic, renal, or gastrointestinal diseases or laboratory abnormality.
6. Symptoms or signs of gastrointestinal obstruction requiring parenteral nutrition or hydration or any other gastro-intestinal disorders or abnormalities, including difficulty swallowing, that would interfere with drug absorption.
7. Serious infections in particular if requiring systemic antibiotic (antimicrobial, antifungal) or antiviral therapy, including known hepatitis B and/or C infection and HIV-infection.
8. Symptomatic central nervous system (CNS) metastasis or leptomeningeal carcinomatosis.
9. Known, uncontrolled hypersensitivity to the investigational drugs or their excipients.
10. Hypersensitivity to Nintedanib, peanut or soya, or to any of the excipients of Nintedanib.
11. Significant cardiovascular diseases, including uncontrolled hypertension, clinically relevant cardiac arrhythmia, unstable angina or myocardial infarction within 6 months prior to randomisation, congestive heart failure > NYHA (New York Heart Association) III, severe peripheral vascular disease, clinically significant pericardial effusion.
12. History of major thromboembolic event, such as pulmonary embolism or proximal deep vein thrombosis, unless on stable therapeutic anticoagulation
13. Known inherited predisposition to bleeding or thrombosis.
14. History of a cerebral vascular accident, transient ischemic attack or subarachnoid haemorrhage within the past 6 months.
15. History of clinically significant haemorrhage in the past 6 months.
16. Major injuries or surgery within the past 28 days prior to start of study treatment or planned surgery during the on-treatment study period.
17. Pregnancy or breastfeeding. Patients with preserved reproductive capacity must have a negative pregnancy test (β-HCG test in urine or serum) prior to commencing study treatment.
18. Patients with preserved reproductive capacity, unwilling to use a medically acceptable method of contraception (see section 5.7) for the duration of the trial and for 6 months afterwards.
19. Radiographic evidence of cavitating or necrotic tumours with invasion of adjacent major blood vessels.
20. Any psychological, familial, sociological or geographical consideration potentially hampering compliance with the study protocol and follow up schedule; those considerations should be discussed with the patient before registration in the trial.
21. Patients who have already received maximal lifetime dose of anthracycline or have experienced cardiac toxicity from an anthracycline should not receive doxorubicin or Paclitaxel Liposomal Doxorubicin (PLD).

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2015-04; Primary Completion 2020-03 (Estimated); Study Completion 2021-03 (Estimated)

PRIMARY OUTCOMES:
Progression Free Survival (PFS) | from date of randomisation to date of progression or death, which ever occurs earlier. Assessed up to 5 years 3 months
  To estimate the progression free survival (PFS) in women with relapsed clear cell carcinoma of the ovary, peritoneum or fallopian tube treated with Nintedanib and compare this to PFS in women treated with chemotherapy.

SECONDARY OUTCOMES:
Overall Survival | defined as the number of days from date of randomisation to date of death (irrespective of reason). Assessed up to 5 years 3 months
  To estimate overall survival in women with relapsed clear cell carcinoma of the ovary, peritoneum or fallopian tube treated with Nintedanib and compare this to OS in women treated with chemotherapy.
Disease control rate | 12 weeks
  Disease control rate (Complete response, partial response and stable disease) at 12 weeks
Quality of Life (QoL) | up to 5 years
  Measured by EORTC QLQ C30 (EORTC Quality of Life Questionnaire Core 30) questionnaire. To assess quality of life in women with relapsed clear cell carcinoma of the ovary, peritoneum or fallopian tube and endometrium treated with Nintedanib and compare this to women treated with chemotherapy.
Quality of Life (QoL) | up to 5 years
  Measured by EORTC OV28 (Ovarian Cancer Module) questionnaire. To assess quality of life in women with relapsed clear cell carcinoma of the ovary, peritoneum or fallopian tube and endometrium treated with Nintedanib and compare this to women treated with chemotherapy.
Quality of Life - recent symptoms of disease and treatment | up to 5 years
  Measured by (Measure of Ovarian Cancer Symptoms and Treatment Concerns) MOST - Recent questionnaire. To measure recent symptoms of disease and treatment in women with relapsed clear cell carcinoma of the ovary, peritoneum or fallopian tube and endometrium treated with Nintedanib and compare this to women treated with chemotherapy.
Q-TWIST (Quality-Adjusted Time Without Symptoms of Disease or Toxicity of Treatment) | up to 5 years
  Measured by EuroQol Group questionnaire EQ-5D. Q-TWiST (Quality-Adjusted Time Without Symptoms of Disease or Toxicity of Treatment) will balance quality and quantity of time by combining survival data with EQ-5D quality of life data. Periods of time spent in ill health due to treatment toxicity or disease symptoms are weighted by average EQ-5D to give a quality of life adjusted time which is combined with a similarly adjusted time spent without either toxicity or symptoms
Response Rate | up to 2 years
  To estimate response rate (RR) in women with relapsed clear cell carcinoma of the endometrium treated with Nintedanib and those treated with chemotherapy. Best response rate will be determined according to a combined GCIG criteria and RECIST criteria Version 1.1
Toxicity | median 12 months
  Adverse event data will be collected during the treatment phase of the study. This will be coded and graded as per NCI-CTCAE v4.0. At the end of treatment, all patients presenting with grade 2 or above toxicities are assessed every 4 weeks until resolution of the toxicity or until another cancer treatment is administered.

CONTACTS AND LOCATIONS:
Overall Officials: Rosalind Glasspool, Principal Investigator — NHS Greater Glasgow and Clyde
Locations (17):
- United Kingdom (17):
  - Beatson West of Scotland Cancer Centre, Glasgow, Lanarkshire
  - Ninewells Hospital, Dundee, Tayside
  - Clatterbridge Cancer Centre, Liverpool, Wirral
  - Belfast City Hospital (Northern Ireland Cancer Centre), Belfast
  - Bristol Heamatology and Cancer Centre, Bristol
  - Velindre Hospital, Cardiff
  - Kent & Canterbury Hospital, Kent
  - Queen Elizabeth Queen Mother Hospital, Kent
  - William Harvey Hospital, Kent
  - St James Hospital, Leeds
  - Guy's Hosital, London
  - Royal Marsden Hospital, London
  - St Bartholomew's Hospital, London
  - University College London Hospital, London
  - The Christie Hospital, Manchester
  - Great Western Hospital, Swindon
  - Musgrove Park Hospital, Taunton

IPD SHARING:
Plan to Share IPD: Yes
It is proposed that data generated by the study will be available 2 years after completion of the trial, or after publication of the first major paper describing the dataset, whichever occurs sooner.

REFERENCES:
- [Derived] Gaitskell K, Rogozinska E, Platt S, Chen Y, Abd El Aziz M, Tattersall A, Morrison J. Angiogenesis inhibitors for the treatment of epithelial ovarian cancer. Cochrane Database Syst Rev. 2023 Apr 18;4(4):CD007930. doi: 10.1002/14651858.CD007930.pub3. PMID 37185961